CLINICAL TRIAL: NCT06188377
Title: Application of Bioimpedance Vector Analysis in Neonates
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-KY-154
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2023-11

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: measured by a impedance analyzer — the healthy chinese neonates will be measured by a impedance analyzer, and will be compared with that of other ethnicity whose data have been reported by literatures.

SUMMARY:
The goal of this observational study is to learn about the distribution of bioimpedance vector of healthy neonates in China in health conditions. The main question it aims to answer are:whether the distribution of bioimpedance vector of healthy neonates in China is correspond to that in other countries.Participants will be measures by NUTRILAB impedance analyzer (Akern, Florence, Italy).

DETAILED DESCRIPTION:
Data such as demographic data, maternal background, gestational age at birth, gestational history, weight and height, will be collected from medical records.Each day we will measure 3 newborns chosen by simple random sampling, for which we will use Excel function.Bioimpedance analysis will be performed according to the manufacturer's instructions within the first 24 hours of life, using a tetrapolar configuration of electrodes (at 400 μA and 50 kHz) with a NUTRILAB impedance analyzer (Akern, Florence, Italy). BIA data will be acquired when they are still, preferably in quiet sleep, avoiding contact between the upper limbs and trunk, and between the legs. Two outer distal adhesive electrodes will be placed on the dorsal surface of the right hand and foot, proximal to the metacarpal-phalangeal and metatarsal-phalangeal joints, and 2 inner electrodes will be placed proximally on the right fore-arm and pretibial region, leaving 5.5cm of free skin around the outer electrodes. The surface should have no skin lesions and will be cleaned with chlorhexidine solution. R and Xc values will be measured in triplicate in each infant, and the arithmetic mean will be used. The device will be calibrated every 20 evaluations(approximately once a week) using a resistor provided by the manufacturer. All the measurements will be performed at the nursery by the same investigator.We will use BIVA to analyse the result: the components of the impedance vector (R and Xc) will be normalized by the height (R/H [ohm/m] and Xc/H [ohm/m], respectively). PA is obtained from the arc-tangent ratio Xc:R. To transform it from radians to degrees, the result is multiplied by 180°/π。Using the RXc graph method the bivariate 95% confidence intervals (ellipses) of the mean vectors of the newborns will be established. From the bivariate normal distribution of R/H and Xc/H, the bivariate 95%, 75%, and 50% tolerance intervals will be drawn. We will use the Hotelling T2 test and univariate analysis (F test) by the BIVA software 2002 for the analysis of the CI for the comparison of the subject groups and for the analysis of tolerance intervals. The significance level is set at 0.05 in all tests.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy term neonates of both sexes within 24 hours.
2. Neonates whose parents or guardians consent with the research.

Exclusion Criteria:

1. Infants with some disease and conditions that could interfere in the body composition (such as heart failure, blue light irradiation, sepsis, kidney injury, hepatic failure, transfusion) and newborns with congenital anomalies and/or genetic problems.
2. Neonates whose parents or guardians refuse to participate in the research.

Max Age: 24 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Chinese healthy term newborns born within 24 hours.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
the distribution of bioimpedance vector of chinese neonates | till 2023-11-30
  collect resistance and reactance of the subjects

CONTACTS AND LOCATIONS:
Overall Officials: Wang Bin, Doctor, Study Director — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Piccoli A, Fanos V, Peruzzi L, Schena S, Pizzini C, Borgione S, Bertino E, Chiaffoni G, Coppo R, Tato L. Reference values of the bioelectrical impedance vector in neonates in the first week after birth. Nutrition. 2002 May;18(5):383-7. doi: 10.1016/s0899-9007(02)00795-5. PMID 11985941
- [Result] Savino F, Grasso G, Cresi F, Oggero R, Silvestro L. Bioelectrical impedance vector distribution in the first year of life. Nutrition. 2003 Jun;19(6):492-6. doi: 10.1016/s0899-9007(02)00947-4. PMID 12781847
- [Result] Toffano RBD, Hillesheim E, Margutti AVB, Camelo Junior JS, Ferraz IS, Del Ciampo LA, Monteiro JP. Bioelectrical Impedance Vector Analysis in Healthy Term Infants in the First Three Months of Life in Brazil. J Am Coll Nutr. 2018 Feb;37(2):93-98. doi: 10.1080/07315724.2017.1364678. Epub 2017 Nov 7. PMID 29111907
- [Result] Margutti AV, Monteiro JP, Camelo JS Jr. Reference distribution of the bioelectrical impedance vector in healthy term newborns. Br J Nutr. 2010 Nov;104(10):1508-13. doi: 10.1017/S000711451000245X. Epub 2010 Jul 2. PMID 20594393